CLINICAL TRIAL: NCT03853837
Title: Ventricular and Pulmonary Vascular Reserve After the Fontan Operation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Other Study IDs: 17-010090; 1K23HL141448-01 (NIH)
Record Dates: First submitted 2018-08-09; First posted 2019-02-26 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Congenital Heart Disease
MeSH Terms: conditions — Heart Failure; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Fontan patients: Fontan patients to be enrolled and complete study tests/procedures
  Interventions: Diagnostic Test: rest-exercise echocardiography
- Retrospective Fontan patients: Fontan patients to be retrospectively reviewed and used as control subjects

INTERVENTIONS:
Diagnostic Test: rest-exercise echocardiography — an echocardiogram performed during rest and exercise
  Groups: Prospective Fontan patients

SUMMARY:
Aim #1: Define and determine the prevalence of pulmonary vascular disease and diastolic dysfunction as assessed by the gold standard of invasive hemodynamic cardiopulmonary exercise testing.

Aim #2: Determine the role of rest-exercise echocardiography for the assessment hemodynamics in Fontan physiology.

Aim #3: Evaluate the clinical impact of pulmonary vascular disease and ventricular diastolic dysfunction.

DETAILED DESCRIPTION:
Define and determine the prevalence of pulmonary vascular disease and diastolic dysfunction as assessed by the gold standard of invasive hemodynamic cardiopulmonary exercise testing. Subjects with Fontan palliation will undergo cardiac catheterization during exercise. The investigators hypothesize that invasive hemodynamic assessment during supine exercise will enable identification of early stage pulmonary vascular disease and diastolic dysfunction that is not apparent from invasive studies performed at rest.

Determine the role of rest-exercise echocardiography for the assessment hemodynamics in Fontan physiology. Transthoracic echocardiography will be performed at rest and during exercise simultaneously with catheterization in the subjects participating in Aim #1 to determine correlations between invasive and noninvasive hemodynamics and identify noninvasive alternatives to assess functional reserve.

Evaluate the clinical impact of pulmonary vascular disease and ventricular diastolic dysfunction. Multi-organ function and patient reported outcomes will be evaluated at baseline, 12 months (optional), and 24 months (optional) in subjects participating in Aims #1 and #2. The investigators hypothesize that subjects with poorer ventricular-vascular reserve will display more clinical and end-organ deterioration in longitudinal follow up.

ELIGIBILITY:
Inclusion Criteria:

* Fontan Palliation
* Age ≥18 years

Exclusion Criteria:

-No clinical indication for cardiac catheterization

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fontan palliation
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Fontan Associated Liver Disease | 5 year
  Fontan associated liver disease measured via magnetic resonance elastography to find liver stiffness measured in kiloPascals:
  <2.5kPa = Normal; 2.5 to 3.0 kPa = Normal or inflammation; 3.0 to 3.5 kPa = Stage 1-2 fibrosis; 3.5 to 4 kPa = Stage 2-3 fibrosis; 4 to 5 kPa = Stage 3-4 fibrosis; >5 kPa = Stage 4 fibrosis;

SECONDARY OUTCOMES:
Mortality | 5 years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials